CLINICAL TRIAL: NCT02155140
Title: Randomised Trial of Enteral Feeding in Patients Discharged From Hospital Following Surgical Resection of an Upper Gastrointestinal Malignancy
Brief Title: Enteral Feeding in Discharged Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to recruit full number of patients
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R&D 11/P/022; 10/H0106/80 (Other: National Research Ethics Service)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Surgical Resection of an Upper Gastrointestinal Malignancy; Nutritional Supplementation Via a Jejunostomy Post Discharge From Hospital
Keywords: enteral feeding; Discharged; surgical resection of an upper gastrointestinal malignancy; Nutritional supplementation via a jejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jejunal feeding (Active Comparator): Nutritional supplementation via their jejunostomies for six weeks post hospital discharge, with continued assessment for a further 18 weeks.
  Interventions: Dietary Supplement: Jejunal feeding
- No jejunal feeding (No Intervention): No jejunal feeding of patients for six weeks following hospital discharge, with continued assessment for a further 18 weeks

INTERVENTIONS:
Dietary Supplement: Jejunal feeding — A feeding jejunostomy tube is inserted at the time of surgery to provide enteral nutritional support.
  Arms: Jejunal feeding

SUMMARY:
Patients due to undergo surgery for oesophageal and gastric malignancy are often malnourished. Up to 10% of patients preoperative weight may also be lost during the early postoperative period. Following discharge from hospital the mechanics of the surgery leads to a loss of gastric reservoir function, lack of appetite, altered intestinal motility and gastro-oesophageal reflux which usually results in reduced dietary intake and further weight loss. In patients who have undergone upper gastrointestinal resections there are no studies examining the benefit of nutritional supplementation following hospital discharge, however, studies in other groups of surgical patients have failed to show benefit. Despite patients who have undergone upper gastrointestinal surgery being 'at risk' nutritionally, there is no evidence demonstrating the value or not of nutritional supplementation following hospital discharge.

Hypothesis: The postoperative under nutrition seen after upper gastrointestinal surgery will exacerbate the reduced quality of life and fatigue patients' already experience. The investigators hypothesise that improving patient's nutritional intake following hospital discharge will improve their quality of life and fatigue levels.

DETAILED DESCRIPTION:
For patients undergoing upper gastrointestinal (GI) surgery for cancer:

1. Because of the nature of upper gastrointestinal surgery these patients have been shown to suffer undernutrition and weight loss after hospital discharge (up to 3 months) and to a greater extent than other groups of surgical patients. Quality of life and fatigue is a major issue after upper GI surgery.
2. Nutritional supplementation via a jejunostomy after hospital discharge is only done routinely for all patients in 10%, and for selected patients in 20% of United Kingdom (UK) hospitals.
3. Derriford hospital is very unusual in that 85% of patients are given home jejunal feeding.
4. In Devon and Cornwall home enteral nutrition is delivered under contract by Fresenius Kabil (a global health care company).
5. There are no studies of home nutritional supplementation in upper GI surgical patients.
6. Studies of home nutritional supplementation in surgical patients having undergone colorectal surgery have not shown clinical or Quality of Life (QoL) benefit despite weight gain.
7. The process of enteral nutrition may be associated with a reduction in quality of life.
8. There is a need for a clinical trial to establish the benefit of home enteral nutritional supplementation. The results of any such trial may influence the highly variable nutritional present practice and may influence the surgeons desire to place a feeding jejunostomy (or not) at surgery which is associated with clinical complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give written informed consent,
* Have had a feeding jejunostomy placed at surgery,
* Competent (or their carer) to set up and use the jejunostomy feeding apparatus themselves.

Exclusion Criteria:

* Participating in another interventional trial,
* Age <18,
* Pre-operative BMI > 35,
* Pre-operative BMI <18,
* Oral intake at hospital discharge of > 90% of requirements,
* It is felt that they or their carers would not to cope with home tube feeding Patients unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Fatigue | 18 weeks
  The primary outcome will therefore be fatigue as measured by the multidimensional fatigue inventory (MFI-20) score. The MFI-20 is divided into five scales: general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue.

SECONDARY OUTCOMES:
Quality of life | 18 weeks
  We will use the oesophagus specific quality of life (QLQ-OES18) scale. The QLQ-OES18 scale is a disease specific Health-related quality of life (HRQL) questionnaire, designed to examine the influence of upper gastrointestinal pathology on patients and improvement in HRQL following treatment.
Health economic analysis | 18 weeks
  Health economic analysis will be based on the EuroQol (EQ 5D) scale 4 (this scale defines health in terms of five dimensions: mobility, self care, usual activities, pain and anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Lewis, MBBS, MD, Study Director — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom